CLINICAL TRIAL: NCT04323865
Title: Non-invasive Fetal Electrocardiography (NI-FECG); Repeatability of Time-domain and Spectral Analyses
Brief Title: Fetal Heart Rate Variability
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); Hartmann Fonden (Other); Augustinus Fonden (Other); The Dagmar Marshall Foundation (Other); AP Moeller Foundation (Other); Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: fHRV_1
Record Dates: First submitted 2020-02-20; First posted 2020-03-27 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-02

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study 2. Repeatability of FHRV
  Interventions: Diagnostic Test: fetal heart rate variability

INTERVENTIONS:
Diagnostic Test: fetal heart rate variability — No direct intervention, as the study is observational.

SUMMARY:
Need statement

- a new way to distinguish between a healthy small fetus and a small fetus suffering from deprivation of nutrition and oxygen to prevent unnecessary induction of preterm birth and improve neonatal outcome.

Aim - to characterize fetal heart rate variability (fHRV) based on fetal ECG in the normal fetus and in the fetus suffering from growth retardation to evaluate its value and applicability as a supplementary tool in fetal surveillance.

Aim of current study

- To evaluate the feasibility of NI-FECG from gestational week 20 and onwards and investigate if important factors as length and heart rate pattern affects repeatability of time domain and spectral analyses in fetuses.

ELIGIBILITY:
Inclusion Criteria:

• Healthy singleton pregnancies

Exclusion Criteria:

• Fetal malformations, multiple pregnancy, obstetric complications, maternal chronic disease and labor.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Danish. Healthy. Pregnant women. Expecting a healthy fetus.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Standard deviation of normal to normal RR-interval (SDNN) | 01.04.2020
  Time domain analysis, measured in ms
Root mean square of successive RR-interval differences (RMSSD) | 01.04.2020
  Time domain analysis, measured in ms
Low frequency power (LF-power) | 01.04.2020
  Spectral analysis, measured in ms^2
High frequency power (HF-power) | 01.04.2020
  Spectral analysis, measured in ms^2
LF-power/HF-power | 01.04.2020
  Spectral analysis, ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Arhus Universityhospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No